CLINICAL TRIAL: NCT01311024
Title: Indirect Effects of Pneumococcal Vaccine on Nasopharyngeal Carriage: a FinIP Effectiveness Trial Satellite Study
Brief Title: Indirect Effects of Pneumococcal Vaccine on Nasopharyngeal Carriage
Acronym: FinIPcarr
Status: Completed | Type: Observational
Sponsor: Arto Palmu (Other Government)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Arto Palmu, Head of Clinical Research Unit, Finnish Institute for Health and Welfare
Organization: Finnish Institute for Health and Welfare (Other Government)
Other Study IDs: THL/1843/6.02.01/2010
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Pneumococcal Infections
Keywords: Children; Pneumococcal Vaccines
MeSH Terms: conditions — Pneumococcal Infections | interventions — twinrix; Hepatitis B Vaccines; Vaccines; Hepatitis A Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Nasopharyngeal and oropharyngeal swabs obtained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sibling vaccinated with PCV GSK1024850A: Older sibling of a child vaccinated with Pneumococcal conjugate vaccine GSK1024850A in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380)
  NOTE: the primary analysis cohort include siblings of the PCV-vaccinated according to infant schedules (excluding siblings of catch-up vaccinated children)
  Interventions: Biological: PCV GSK1024850A
- Control-vaccinated sibling: Older sibling of a child vaccinated with control vaccine (hepatitis B vaccine or hepatitis A vaccine) in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380)
  NOTE: the primary analysis cohort include siblings of the PCV-vaccinated according to infant schedules (excluding siblings of catch-up vaccinated children)
  Interventions: Biological: hepatitis B vaccine or hepatitis A vaccine

INTERVENTIONS:
Biological: PCV GSK1024850A — 2 to 4 doses administered to the siblings in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380)
  Other Names: GSK Biologicals' Synflorix TM vaccine
  Groups: Sibling vaccinated with PCV GSK1024850A
Biological: hepatitis B vaccine or hepatitis A vaccine — 2 to 4 doses administered to the siblings in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380)
  Other Names: GSK Biologicals' Engerix TM (hepatitis B) vaccine; GSK Biologicals' Havrix TM (hepatitis A) vaccine
  Groups: Control-vaccinated sibling

SUMMARY:
The purpose of this study is to assess the indirect effects of a pneumococcal conjugate vaccine administered to infants on vaccinees' elder non-vaccinated siblings aged 3 to 7 years.

DETAILED DESCRIPTION:
The purpose of this study is to assess the indirect effects of a pneumococcal conjugate vaccine administered to infants on vaccinees' elder non-vaccinated siblings aged 3 to 7 years.

This study includes a cross-sectional sampling of nasopharyngeal and oropharyngeal swabs in 2011 and a register-based follow-up study for invasive disease, hospital-diagnosed pneumonia, tympanostomy tube surgery and outpatient antimicrobial treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 3 to 7 years
* younger sibling at least 12 months of age living in the same household participates in the FinIP or 053 trial (regardless of the vaccination schedule)
* at least one parent with fluent Finnish
* informed consent from one parent

Exclusion Criteria:

* commercial PCV vaccination administered
* study-related PCV vaccination administered (open or blind)
* history of antimicrobial treatment within 4 weeks (the child can be enrolled later)

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Non-PCV-vaccinated 3 to 7 year-old siblings living in the same household with a younger child vaccinated in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380)
Sampling Method: Non-Probability Sample
Enrollment: 2341 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arto A Palmu, M.D., Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- National Institute for Health and Welfare, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Public webpage for the FinIP trial and the carriage study — http://www.finip.fi

RESULTS

PARTICIPANT FLOW:
Groups:
- PCV-vaccinated Sibling (GSK1024850A): Older sibling of a child vaccinated with PCV in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380)
  Pneumococcal conjugate vaccine GSK1024850A: 2 to 4 doses administered to the siblings in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380).
  Evaluable subjects with NPS sample analysed 482 Siblings of infant-vaccinated children in the PCV 2+1 arm and 445 Siblings of infant-vaccinated children in the PCV 3+1 arm and 568 Siblings of catch-up vaccinated children in the PCV arms 1495 in total
- Control-vaccinated Sibling: Older sibling of a child vaccinated with control vaccine (hepatitis B vaccine or hepatitis A vaccine) in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380)
  hepatitis B vaccine or hepatitis A vaccine: 2 to 4 doses administered to the siblings in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380)
  Evaluable subjects with NPS sample analysed 518 Siblings of infant-vaccinated children in the control arms and 271 Siblings of catch-up vaccinated children 789 in total
Period: Overall Study
Arm/Group | PCV-vaccinated Sibling (GSK1024850A) | Control-vaccinated Sibling
Started | 1530 | 811
Completed | 1495 | 789
Not Completed | 35 | 22
Not completed — Protocol Violation | 35 | 22

BASELINE CHARACTERISTICS:
Population: These numbers include only the siblings of the infant-vaccinated FinIP children.
Groups:
- PCV-vaccinated Sibling (GSK1024850A): Older sibling of a child vaccinated with PCV in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380)
  Pneumococcal conjugate vaccine GSK1024850A: 2 to 4 doses administered to the siblings in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380)
- Control-vaccinated Sibling: Older sibling of a child vaccinated with control vaccine (hepatitis B vaccine or hepatitis A vaccine) in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380)
  hepatitis B vaccine or hepatitis A vaccine: 2 to 4 doses administered to the siblings in the cluster-randomized Finnish Invasive pneumococcal Disease Trial (ClinicalTrials.gov Identifier:NCT00861380)
- Total: Total of all reporting groups
Arm/Group | PCV-vaccinated Sibling (GSK1024850A) | Control-vaccinated Sibling | Total
Number analyzed (Participants) | 927 | 518 | 1445
Age, Continuous [Median (Full Range); unit: years] | 4 [3 to 7] | 4 [3 to 7] | 4 [3 to 7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 468 | 257 | 725
  Male | 459 | 261 | 720

OUTCOME MEASURES:

1. Primary Outcome: Carriage Due to Any Pneumococcal Serotype Included in the Ten-valent Pneumococcal Conjugate Vaccine (PCV10) Vaccine in Older Siblings of Children Vaccinated With Infant Schedules
Description: Carriage due to any pneumococcal serotype included in the ten-valent pneumococcal conjugate vaccine (PCV10) vaccine in older siblings of children vaccinated with infant schedules. Nasopharyngeal swabs taken once at 3 to 7 years of age when the vaccinated sibling is at least 12 months of age
Time Frame: one sampling at 3 to 7 years of age
Measure: Number; unit: percentage of subjects
Arm/Group | PCV-vaccinated Sibling (GSK1024850A) | Control-vaccinated Sibling
Number analyzed (Participants) | 927 | 518
percentage of subjects | 14.5 | 19.3

2. Secondary Outcome: Carriage Due to Any Pneumococcal Serotype
Description: Nasopharyngeal and oropharyngeal swabs taken once at 3 to 7 years of age when the vaccinated sibling is at least 12 months of age
Time Frame: one sampling at 3 to 7 years of age
Reporting Status: Not Posted

3. Secondary Outcome: Carriage Due to Haemophilus Influenzae
Description: as for outcome 2
Time Frame: one sampling at 3 to 7 years of age
Reporting Status: Not Posted

4. Secondary Outcome: Invasive Pneumococcal Disease
Description: Register follow-up up to 8 years after the vaccination of the younger sibling in the family
Time Frame: Up to 8 years
Reporting Status: Not Posted

5. Secondary Outcome: Hospital-diagnosed Pneumonia
Description: Register follow-up up to 8 years after the vaccination of the younger sibling in the family
Time Frame: Up to 8 years
Reporting Status: Not Posted

6. Secondary Outcome: Tympanostomy Tube Surgery
Description: Register follow-up up to 8 years after the vaccination of the younger sibling in the family
Time Frame: Up to 8 years
Reporting Status: Not Posted

7. Secondary Outcome: Outpatient Antibiotic Treatment
Description: Register follow-up up to 8 years after the vaccination of the younger sibling in the family
Time Frame: Up to 8 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Study-related adverse events collected, i.e. those due to NPS and OPS sampling.
Description: Note, this study did not include active vaccination of the participants, but indirect impact of the vaccination given to younger siblings was evaluated.
Arm/Group | PCV-vaccinated Sibling (GSK1024850A) | Control-vaccinated Sibling
Serious Adverse Events (participants affected / at risk) | 0/1495 | 0/789
Other Adverse Events (participants affected / at risk) | 0/1495 | 0/789

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No